CLINICAL TRIAL: NCT03491826
Title: Fetal and Maternal Outcome in Preterm Premature Rupture of Membranes (PPROM) at AIN Shams Maternity Hospital: A Retrospective Analysis of Last Five Years Admissions
Brief Title: Fetal and Maternal Outcome in Preterm Premature Rupture of Membranes (PPROM)
Status: Completed | Type: Observational
Sponsor: sarah mohamed hassan (Other)
Collaborators: Hend Mostafa Hussein Salem (Unknown)
Responsible Party: Sponsor-Investigator, sarah mohamed hassan, lecturer of obstetrics and gynecology, Kasr El Aini Hospital
Organization: Kasr El Aini Hospital (Other)
Other Study IDs: 123
Record Dates: First submitted 2018-03-28; First posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Premature Rupture of Membrane
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ROM before 34 weeks (A): premature rupture of membrane before 34 weeks
  Interventions: Biological: rupture of membrane
- ROM after 34 weeks (B): premature rupture of membrane after 34 weeks
  Interventions: Biological: rupture of membrane

INTERVENTIONS:
Biological: rupture of membrane

SUMMARY:
The aim of this study is to compare fetal and maternal outcome in cases of PPROM before 34 weeks versus after 34 weeks.

DETAILED DESCRIPTION:
The data will be retrieved from the archival files and analyzed

ELIGIBILITY:
Inclusion Criteria:

* rupture of membrane

Exclusion Criteria:

* medical disorder

Ages: 24 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant female with history of rupture membrane
Sampling Method: Probability Sample
Enrollment: 1011 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
maternal mortality | up to 48 hours after delivery
  maternal mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainiy Hospital, Cairo, Egypt